CLINICAL TRIAL: NCT06393309
Title: Investigation of Long-term Outcome of Levetiracetam and Valproate in Treatment of Idiopathic Generalized Epilepsy
Brief Title: Levetiracetam Versus Valproate in Idiopathic Generalized Epilepsy
Acronym: LEVAGE
Status: Completed | Type: Observational
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Associate professor of neurology, Mazandaran University of Medical Sciences
Other Study IDs: 14751
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Treatment of Idiopathic Generalized Epilepsy
Keywords: Levetiracetam; Valproate; Idiopathic generalized epilepsy
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized | interventions — Levetiracetam; Valproic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Levetiracetam: Patients with idiopathic generalized epilepsy who were under treatment with levetiracetam
  Interventions: Drug: Levetiracetam
- Sodium valproate: Patients with idiopathic generalized epilepsy who were under treatment with valproate
  Interventions: Drug: Sodium valproate

INTERVENTIONS:
Drug: Levetiracetam — Patients with idiopathic generalized epilepsy who were under treatment with levetiracetam
  Groups: Levetiracetam
Drug: Sodium valproate — Patients with idiopathic generalized epilepsy who were under treatment with valproate
  Groups: Sodium valproate

SUMMARY:
This study aimed to compare the long-term efficacy and safety of levetiracetam and valproate in treatment of idiopathic generalized epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of juvenile myoclonic epilepsy or generalized tonic-clonic seizure alone
* Regular monotherapy with levetiracetam or sodium valproate

Exclusion Criteria:

* Poor drug adherence
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with idiopathic generalized epilepsy (juvenile myoclonic epilepsy or generalized tonic-clonic seizure alone) who are on monotherapy with levetiracetam or sodium valproate
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Seizure free rate | 1 to 5 years
  The percent of patients who remained seizure free on treatment
Time to first seizure | 1 to 5 years
  The interval between start of treatment and recurrence of seizure

SECONDARY OUTCOMES:
Retention rate | 1 to 5 years
  The percent of patients who remained on treatment with levetiracetam or valproate
Time to withdrawal | 1 to 5 years
  The interval between start and withdrawal of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bu Ali Sina Hospital, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: No